CLINICAL TRIAL: NCT06476990
Title: Food Rx + CHW: a Community Health Worker-led Medically Tailored Grocery Intervention to Address Food Insecurity and Type 2 Diabetes
Brief Title: Food Rx + Community Health Worker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Principal Investigator, Kristina Bridges, Research Assistant Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00144654
Record Dates: First submitted 2024-06-20; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food-only group (Active Comparator)
  Interventions: Behavioral: Healthy food box
- Food + CHW group (Experimental)
  Interventions: Behavioral: Healthy food box

INTERVENTIONS:
Behavioral: Healthy food box — All participants received 12 weekly deliveries of food containing approximately $8 worth of shelf-stable food items purchased from a local food bank (beans, canned vegetables and no-sugar added fruit, shelf-stable dairy products, canned tuna, and whole grains) and $25 of fresh produce (5-7 items including leafy greens, peppers, potatoes, broccoli, carrots, zucchini, cauliflower, celery, cabbage, asparagus, apples, or strawberries). When seasonably available, fresh vegetables and fruit were sourced from local farmers via a local food hub. In addition to food, participants in the Food + CHW group also received 7 weekly virtual sessions with a CHW (four 90-minute ZOOM counseling sessions and three 30 to 60-minute check-in phone calls). CHW sessions included diabetes-appropriate cooking and nutrition education and personalized benefit enrollment and linkage to existing food access resources (for example SNAP, Double up Food Bucks, and Kansas Senior Farmers Market Vouchers).
  Other Names: Community health worker

SUMMARY:
Food insecurity increases an individual's risk of poor health outcomes from some of the most costly and preventable chronic diseases, including type 2 diabetes. The goal of this interventional pilot study is to see if primary care patients with self-reported food insecurity and a diagnosis of type 2 diabetes who receive 12 weekly home deliveries of fresh produce and diabetes-appropriate, shelf-stable food will have improved diabetes management. Half of these patients also received support from a community health worker (CHW) including nutrition and cooking education and tailored assistance accessing food resources and other social needs (example: transportation). The investigators hypothesized that participants receiving support from a CHW along with food boxes would have greater improvement in health outcomes compared to those participants who received only food.

DETAILED DESCRIPTION:
Food Rx + CHW is a 3-month community health worker led medically tailored grocery intervention for patients with self-reported food insecurity and a diagnosis of type 2 diabetes at one academic medical center in the Midwest United States. Prior to contact and recruitment, eligible patients were randomly assigned to receive 12 weekly food deliveries and support from a CHW (Food + CHW group) or food deliveries only (Food-only group).

All participants receive 12 weekly contactless deliveries of food. CHWs conduct three virtual study visits with participants to administer surveys and/or collect biomarker measurements at weeks 1, 12, and 24. No changes in the frequency of visits with the patient's provider are recommended. Virtual visit 1 involves the completion of study forms, assessment of household size for most meals, cultural preferences, food allergies, baseline cooking and eating habits, and assessment for knowledge and usage of local and/or federal food support programs. At week 12, participants use at home kits and devices (provided by the study) to measure and report their HbA1C, weight and blood pressure and complete post-intervention surveys on diet, knowledge and usage of food access programs and resources, and an anonymous feedback questionnaire on the strengths and opportunities for improvement in the program. At week 24, participants measured and reported their final HbA1C, weight and self-collected blood pressure result.

In addition to food, participants in the Food + CHW group also received 7 weekly virtual sessions with a CHW (four 90-minute ZOOM counseling sessions and three 30 to 60-minute check-in phone calls). CHW sessions included diabetes-appropriate cooking and nutrition education and personalized benefit enrollment and linkage to existing food access resources (for example Supplemental Nutrition Assistance Program, Double up Food Bucks, and Kansas Senior Farmers Market Vouchers).

Each weekly food box contained approximately $8 worth of shelf-stable food items purchased from a local food bank (beans, canned vegetables and no-sugar added fruit, shelf-stable dairy products, canned tuna, and whole grains) and $25 of fresh produce (5-7 items including leafy greens, peppers, potatoes, broccoli, carrots, zucchini, cauliflower, celery, cabbage, asparagus, apples, or strawberries). When seasonably available, fresh vegetables and fruit were sourced from local farmers via a local food hub. When local produce was not available, CHWs sourced produce from grocery stores.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking,
* Diagnosis of type 2 diabetes with a most recent HbA1C > 7,
* Previously answered "yes" to the food insecurity needs question ("In the last 12 months, did you ever eat less than you should because there wasn't enough money for food?") on a SDOH screener during a patient care visit

Exclusion Criteria:

* Participant address was outside the delivery zone (the Kansas City Metro area),
* Participant resides in a facility that provides all meals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average blood glucose, as measured by Hemoglobin A1C | Baseline, 3 months, 6 months
  Hemoglobin A1C point of care test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No